CLINICAL TRIAL: NCT04161950
Title: Prospective Comparison of Two EUS System for Clinical Performance
Brief Title: Assessment of the Echoendoscope for Clinical Performance
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Tao Guo, Associated professor in Department of Gastroenterolgy, Peking Union Medical College Hospital
Other Study IDs: 2017YFC0109804
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Endosonography
Keywords: echoendoscope; endoscopic ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tested device model (EG-UR5-S50 ): Tested device model: The EG-UR5 echoendoscope manufactured by SonoSscope Medical Crop. That used with the HD-500 image processor, HDL-500X light source and S50 ultrasonic processor.
  Interventions: Other: Assessment of the safety and validity of echoendoscope
- Compared device model (GF-UE260-ME2): Compared device model: The GF-UE260 echoendoscope manufactured by Olympus and its compatible light source, image processor and ME2 ultrasonic processor.
  Interventions: Other: Assessment of the safety and validity of echoendoscope

INTERVENTIONS:
Other: Assessment of the safety and validity of echoendoscope — 1. Ultrasonic and endoscopic image quality assessment
  2. Device controllability assessment
  3. System safety assessment
  4. System stability assessment

SUMMARY:
The primary objective for this study is to compare the safety and validity of two endoscopic ultrasonography (EUS) systems (GF-UE260-ME2 and EG-UR5-S50) used for clinical performance and establish a relative EUS performance assessment system and clinical case data to provide support for the product performance improvement.

DETAILED DESCRIPTION:
This research is a random, opening and parallel-controlled clinical test. Tested device model: The EG-UR5 ultrasonic endoscope manufactured by SonoSscope Medical Crop. That used with the HD-500 image processor, HDL-500X light source and S50Exp ultrasonic color doppler instrument .

Compared device model: The GF-UE260-ME2 ultrasonic endoscope manufactured by Olympus and its compatible light source, image processor and ultrasonic instrument.

To scientifically compare the clinical performances of the test model and the compared model, the enrolled objects would be randomly distributed to the tested group and the compared group to conducted the examination with the tested model and the compared model respectively.

EUS will be performed in the standard fashion by one of the experienced endosonographers in the unit. Once the EUS is complete, the procedure will be stopped and the echoendoscope withdrawn from the patient.

1. Check Points Providing optical images of the human upper gastrointesinal tract (including esophagus, stomach and duodenum) for observing, diagnosis and treatment, and for the ultrasonic check and diagnosis for the upper gastrointestinal tract and surrounding organs.
2. Test Items 1. Ultrasonic and endoscopic image quality assessment 2. Device controllability assessment 3. System safety assessment 4. System stability assessment

The data are recorded in the CRF, including patient information, clinical assessment for the usage of the endoscope and device operation, thus to perform a comprehensive assessment whether the safety and validity of this product can meet the clinical requirements.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with clinical indication for the endoscopic ultrasonography examination or diagnosis;
2. Patients volunteering to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Patients do not sign the informed consent.
2. Mental disorders and non-cooperated patient
3. Severe cardiopulmonary diseases (such as severe cardiac dysfunction, severe pulmonary dysfunction and severe arrhythmia)
4. Shock or other severe patient
5. Suspected or confirmed upper digestive tract perforation or perforation acute phase
6. Acute phase of gastric and esophageal chemical burns
7. Patients do not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to PUMCH Endoscopy Unit for EUS assessment will be included.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Ultrasonic Image Quality Assessment | up to 2 months
  Check Points for Ultrasonic Image Esophagus, stomach, cholecyst, bile duct, pancreas and portal vein system Ultrasonic image quality Assessment standards Assess the ultrasonic image quality of all judgment points according to the ranking degree: excellent, well, bad. Only the assessment of all organs are excellent, the ultrasonic image quality is excellent. If one or more than one assessments are good, the ultrasonic image quality is good. If one or more than one assessments are bad, the ultrasonic image quality is bad.
  The comparison of the image qualities of the tested model and compared model is verified by the non-inferior validation method and the boundary is 10%, and the confidence interval rate differential is 95%.
Endoscopic Image Quality Assessment | up to 2 months
  Check Points for endoscopic Image Esophagus, proximal stomach, stomach body,gastric angle,antrum and duodenal bulb.
  Assess the ultrasonic image quality of all judgment points according to the ranking degree: excellent, well, bad. Only the assessment of all observed points are excellent, the endoscopic image quality is excellent. If one or more than one observation points are good, the endoscopic image quality is good. If one or more than one observation points are bad, the endoscopic image quality is bad.
  The comparison of the image qualities of the tested model and compared model is verified by the non-inferior validation method and the boundary is 10%, and the confidence interval rate differential is 95%.

SECONDARY OUTCOMES:
Device controllability Assessment | up to 2 months
  The good ration of the device controllability is computed to assess the performance of the ultrasonic endoscope and the target value is more than 98%.
System safety assessment | up to 2 months
  Judge the device safety according to the system safety adverse events and the target rate (the estimate value) of the events is 0.
System stability assessment | up to 2 months
  Judge the device stability according to the system stability adverse events and the target rate (the estimate value) of the events is less than 5%.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Guo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Gastroenterology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data are private.

REFERENCES:
- [Background] Roubein LB. Endoscopic ultrasonography and the malignant esophageal stricture: implications and complications. Gastrointest Endosc. 1995 Jun;41(6):613-5. doi: 10.1016/s0016-5107(95)70205-9. No abstract available. PMID 7672562
- [Background] Jenssen C, Alvarez-Sanchez MV, Napoleon B, Faiss S. Diagnostic endoscopic ultrasonography: assessment of safety and prevention of complications. World J Gastroenterol. 2012 Sep 14;18(34):4659-76. doi: 10.3748/wjg.v18.i34.4659. PMID 23002335